CLINICAL TRIAL: NCT02880930
Title: Optimizing Vitamin D Status in Children With Pre-school Wheeze or Asthma:a Pilot Study (OPTIVIT)
Brief Title: Optimizing Vitamin D Status in Children With Wheeze / Asthma (OPTIVIT)
Acronym: OPTIVIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 011320
Record Dates: First submitted 2016-08-05; First posted 2016-08-26 (Estimated); Last update posted 2019-04-08 (Actual); Status verified 2018-04

CONDITIONS: Asthmatic Crisis; Wheezing
Keywords: vitamin D
MeSH Terms: conditions — Status Asthmaticus; Respiratory Sounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vitamin D supplement (Cholecalciferol) (Experimental): Participants will be given oral Fultium-D3 drops (Internis) contain 400 IU cholecalciferol/day for a period of 3 months. Daily vitamin D3 supplementation dose will be increased to 1,000 IU for an additional 3 months if plasma 25(OH)D still below 75 nmol/L.
  Interventions: Dietary Supplement: Fultium-D3 drops (Internis)

INTERVENTIONS:
Dietary Supplement: Fultium-D3 drops (Internis) — Oral daily doses of vitamin D3 (400 IU for 3 months; and 1,000 IU for an additional 3 months)

SUMMARY:
Vitamin D deficiency is highly prevalent in the UK. Research shows that vitamin D enhances the immune system and may help protect against chest infections that can cause wheezing illness or worsen asthma symptoms. The Department of Health recommends a dose of 10 micrograms of vitamin D/day to prevent severe vitamin D deficiency in children. However, many studies have reported that this dose is not enough to raise plasma 25(OH)D concentration to the levels most likely to prevent against worsening of asthma symptoms. Such studies suggest that 25 micrograms of vitamin D/day. This dose is safe but its effects on vitamin D blood levels have not yet been specifically tested in children with asthma/wheeze. This study is designed to determine the optimal oral daily vitamin D supplementation dose to treat vitamin D deficiency in children with asthma or preschool wheeze. Over the 6-month course of the study, participants will meet with the study team four times in clinic or in their own home and will be contacted by telephone five times. Children will be asked to give a drop of blood via a fingerprick to test their vitamin D level and a sample of nasal epithelial lining fluid for measurement of inflammatory markers on three separate occasions.

DETAILED DESCRIPTION:
The study is designed to compare the efficacy of a daily oral vitamin D3 supplementation dose of 10 micrograms (400 IU) for 3 months vs a daily oral vitamin D3 supplementation dose of 25 micrograms (1,000 IU) for an additional 3 months in correcting vitamin D deficiency in children with asthma or preschool wheezing illness.

Identification procedures

A member of the patient's usual care team will identify potentially eligible participants from patient records at participating sites. Identified individuals will be contacted by post, giving a brief explanation of the study and asking them to contact a member of the research team if they wish to find out more. A member of the research team will explain the study to them and ask them if they would like to receive the study participant information sheet (PIS). The PIS will be posted to patients expressing an interest in the study; those who subsequently confirm their interest in participation will be re-contacted by the study team, and offered a screening appointment at a study site. Additionally, posters advertising the study and providing contact details for the study team will be displayed in appropriate public places, such as hospital out-patient departments and General Practitioner (GP) surgeries, where potentially eligible participants are likely to see them; advertisements for the study may also be placed in the press, and circulated on email within Queen Mary, University of London. Potentially eligible children who fulfill eligibility criteria and give their assent (if aged ≥7 years) and have consent from their parent/legal guardian will be enrolled in the study.

Study visits

Visit 1 - Screening:

Once the child and their parent/legal guardian decide to take part in the study and sign the agreement forms (assent and consent form), the investigators will record details of children's sociodemographic status, ethnicity, age and sex. The investigators will measure children's body weight and height, and ask children aged >= 5 years to fill in a questionnaire to assess their level of asthma symptom control. The investigators will then collect a drop of each child's blood with a finger-prick to measure his/her vitamin D level and a sample of fluid from one nostril of each child with a small (5 x 25 mm) strip of absorbent material to measure his/her inflammatory status. The investigators will apply a numbing cream or spray to each child's finger before the fingerprick to minimise discomfort.

Telephone contact T1:

The investigators will telephone children's parents/legal guardians to let them know the results of their child's baseline vitamin D test. If this is normal (75 nmol/L or more), then the child does not need a vitamin D supplement: the parent / guardian will be reassured, and the child will not be able to take part in this study. If the level is low, then the investigators will arrange to meet with the child and his/her parent/guardian a second time.

Visit 2 - (1 week later):

At this visit, the investigators will show children's parents/legal guardians how to give their child the study drops each day and also supply them with a bottle of vitamin D drops for their child to take every day at a dose of 6 drops (400 IU; 10 μg) per day. The investigators will also give them a diary where they can record the doses their child takes every day and note down details of unplanned visits to a doctor/nurse due to wheezing illness or worsening of asthma symptoms during the study.

Telephone contact T2 - (One week after Visit 2):

The investigators will telephone parents/legal guardians as arranged to check if their child is taking the study drops and to see how they are getting on. The investigators will also check if their child has made any unplanned visits to a doctor or a nurse due to wheezing illness or worsening of asthma symptoms since the last study visit.

Telephone contact T3 - (Three weeks after telephone call T2):

In this telephone call, the investigators will make the same checks as those in telephone contact T2.

Visit 3 - (Month 3):

In this visit, the investigators will perform the same tests as those in study visit 1. The investigators will take back the bottle with the remaining vitamin D liquid and the completed study diary, and provide a new diary and bottle with study drops.

Telephone contact T4 - (One week after Visit 3):

In this telephone call, the investigators will do the same checks as those in telephone call T2. The investigators will also let parents/legal guardians know results of their child's second vitamin D test. Based on this result, the investigators will decide if their child needs to increase the dose to 15 drops (1,000 IU; 25 μg) per day for a further 3 months or to continue with 6 drops (400 IU; 10 μg) per day for a further 3 months or to stop vitamin D supplementation.

Telephone contact T5 - (Three weeks after telephone call T4):

In this telephone call, the investigators will make the same checks as those in telephone contact T2.

Visit 4 - FINAL VISIT - (Month 6):

In this study visit, the investigators will perform the same tests as those in study visit 1. The investigators will ask parents/legal guardians to complete a final questionnaire about their child's experience in the study. The investigators will take back the bottle with the remaining study drops and the completed study diary. Once enrolment to the study and analysis of all study data is complete, the investigators will write to participants' parents/legal guardians to tell them about our final findings, including results of their child's final vitamin D test.

Additional procedures throughout the study:

Participants' parents/legal guardians will be asked to report the daily supplementation doses their child takes and record details of unplanned healthcare visits to a GP/nurse due to wheezing illness or worsening of asthma symptoms during the study.

If a participant reports symptoms of raised blood calcium level during the study nausea, vomiting or feeling generally unwell), an urgent check of his/her corrected blood calcium level will be performed and an appointment with a pediatrician will be arranged if necessary.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1-12 years

  * For children aged 1-4 years: ≥2 self-reported wheezing illness episodes (as shown in a video recording of a wheeze episode) requiring unscheduled healthcare in the previous year
  * For children aged 5-12 years: doctor diagnosis of asthma and ≥1 self-reported asthma exacerbation requiring an unscheduled healthcare visit in the previous year.
* Children's parent/legal guardian gives informed consent for children.
* If child aged ≥7 years, gives informed assent.

Exclusion Criteria:

* Baseline 25(OH)D concentration ≥75 nmol/L.
* Already taking any vitamin D supplements.
* Any other chronic or recent acute respiratory or systemic condition.
* Already enrolled in another interventional research study

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2016-12; Primary Completion 2019-01 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Proportion of children with vitamin D status above or equal to 75 nmol/L at 3 and 6 months of oral vitamin D3 supplementation | 6 months in total
  Proportion of children with asthma and pre-school wheezing illness with baseline serum 25(OH)D concentration<75 nmol/L attaining serum 25(OH)D concentration >75 nmol/L after 3 months of an oral daily dose of 400 IU and after an additional 3 months of oral daily vitamin D3 supplementation with 1,000 IU

SECONDARY OUTCOMES:
Proportion of children with treatment related adverse events D status at 3 and 6 months of oral vitamin D3 supplementation | 6 months in total
  To define the proportion of individuals with 25(OH)D concentration above 220nmol/L at 3 and 6 months after daily oral vitamin D3 supplementation.
Changes from baseline in concentration of inflammatory mediators in nasal epithelial lining fluid at 3 and 6 months after daily oral vitamin D3 supplementation | 6 months in total
  To determine the effect of different regimens of oral vitamin D supplementation on concentrations of inflammatory mediators in nasal epithelial lining fluid (ELF) at 3 and 6 months
Changes from baseline in childhood Asthma Control Test at 3 and 6 months | 6 months in total
  To determine the difference in childhood asthma control test score (c-ACT) at 3 months vs. 0 months and 6 months vs. 0 months for children ≥5 years.
Adherence to study supplement | 6 months in total
  To determine the proportion of vitamin D3 supplementation doses taken (self-reported and supplement volume assessment) during the study
Capture of unscheduled health care attendances for asthma or wheezing illness (self-reported) | 6 months in total
  To define the number of unscheduled healthcare attendances for asthma exacerbation(s) or wheezing illness as self-reported by individuals and their parents.
Capture of unscheduled health care attendances for asthma or wheezing illness | 6 months in total
  To define the number of unscheduled healthcare attendances for asthma exacerbation(s) or wheezing illness as reported by GP records
Agreement between self-reported and GP record number of unscheduled healthcare visits | 6 months in total
  To evaluate agreement between self-reported and GP record number of unscheduled healthcare attendance for wheezing illness or asthma exacerbation(s).
Determinants of vitamin D status | 6 months in total
  To identify determinants of increase in serum 25(OH)D concentration in response to daily oral vitamin D3 supplementation
Participant's feedback about the study | 6 months in total
  To evaluate children's and parents' experiences of taking part in the study (qualitative evaluation).

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Martineau, Principal Investigator — Barts and The London School of Medicine and Dentistry, Queen Mary University, University of London
Locations (1):
- The Royal London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes